CLINICAL TRIAL: NCT02728427
Title: Multicenter Study on Comparing Suprapubic Catheterization Versus Traditional Transurethral Catheterization in Laparoscopic Surgery for Rectal Cancer
Brief Title: Multicenter Study on Suprapubic Catheterization Versus Transurethral Catheterization in Laparoscopic Surgery for Rectal Cancer
Acronym: MSSPC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Fujian Cancer Hospital (Other Government); Fujian Provincial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SPCCVC-TUC
Record Dates: First submitted 2016-03-22; First posted 2016-04-05 (Estimated); Last update posted 2018-04-26 (Actual); Status verified 2018-04

CONDITIONS: Rectal Cancer; Surgery
Keywords: Suprapubic Catheterization; Transurethral Catheterization; Rectal Cancer; Laparoscopic Surgery
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Suprapubic Catheterization (Experimental): Suprapubic catheterization using central venous catheter(CVC-2 7F) will be performed for patients in this group.
  Interventions: Device: Suprapubic catheterization using central venous catheter(CVC-2 7F)
- Transurethral Catheterization (Active Comparator): Transurethral catheterization using Foley catheter will be performed for patients in this group.
  Interventions: Device: Transurethral catheterization using Foley catheter

INTERVENTIONS:
Device: Suprapubic catheterization using central venous catheter(CVC-2 7F) — Suprapubic catheterization using central venous catheter(CVC-2 7F) will be performed for patients after laparoscopic surgery for rectal cancer.Suprapubic catheterization is inserted at the end of the procedure. It will be clamped depending on surgeon's specific instruction and removed if the urinary residual is less than 50 cc.
  Other Names: SPCCVC
  Arms: Suprapubic Catheterization
Device: Transurethral catheterization using Foley catheter — Traditional transurethral catheterization using Foley catheter will be performed for patients.The catheterization is removed on day 5 in patients without complication.
  Other Names: TUC
  Arms: Transurethral Catheterization

SUMMARY:
Compared with traditional open proctectomy, laparoscopic surgery is associated with less pain, earlier recovery, and better cosmetic outcome, and its long-term oncologic outcomes have been demonstrated. However, the rate of urinary dysfunction after rectal cancer surgery was about 19-38% because of mesorectal excision. The type of drainage is unclear. Some studies show that the rates of urinary tract infection, second catheterization, and urinary symptom are lower with suprapubic catheterization (SPC) than with transurethral catheterization (TUC). Moreover，SPC allows for testing the bladder voiding without drainage removal. Furthermore，SPC using central venous catheter(CVC) is less invasive.

Currently, there is lack of randomized controlled trial(RCT) to compare SPC with TUC. Therefore, investigators perform this prospective randomized trial to compare SPC using CVC with TUC in laparoscopic surgery for rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Pathological rectal carcinoma
* Male patients
* Performance status of 0 or 1 on ECOG (Eastern Cooperative Oncology Group) scale
* ASA (American Society of Anesthesiology) score class I, II, or III
* Laparoscopic surgery for rectal cancer
* Written informed consent

Exclusion Criteria:

* Emergency surgery due to complication (obstruction or perforation) caused by rectal cancer
* Preoperative T4b according to the 7th Edition of AJCC Cancer Staging Manual
* Basic diseases of urinary system (urinary bladder stones and tumors, prostate cancer, neurogenic bladder, urethral stricture) that affect voiding function
* History of previous pelvic surgery
* Severe mental disease

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-04; Primary Completion 2018-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Catherization time | 6 days

SECONDARY OUTCOMES:
Number of catheterization | 30 days
Catheter-Associated Urinary Tract Infection | 30 days
Pain score | 5 days
  Postoperative pain is recorded using the visual analog scale (VAS) pain score tool from the surgery day to the fifth day after surgery.
International Prostatic Symptom Score | 30 days
  The International Prostatic Symptom Score is recorded from the day before surgery to the 30th day after surgery.
Time to first ambulation | 7 days
Duration of hospital stay | 30 days
Urinary extravasation | 30 days
Hematuria | 30 days
Catheter obstruction | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Guoxin Li, M.D., Ph.D., Principal Investigator — Chinese Laparoscopic Gastrointestinal Surgery Study (CLASS) Group; Nanfang Hospital, Southern Medical University, China
Locations (3):
- China (3):
  - Fujian Provincial Hospital, Fuzhou, Fujian
  - Fujian Provincial cancer Hospital, Fuzhou, Fujian
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bonjer HJ, Deijen CL, Abis GA, Cuesta MA, van der Pas MH, de Lange-de Klerk ES, Lacy AM, Bemelman WA, Andersson J, Angenete E, Rosenberg J, Fuerst A, Haglind E; COLOR II Study Group. A randomized trial of laparoscopic versus open surgery for rectal cancer. N Engl J Med. 2015 Apr 2;372(14):1324-32. doi: 10.1056/NEJMoa1414882. PMID 25830422
- [Background] Jayne DG, Brown JM, Thorpe H, Walker J, Quirke P, Guillou PJ. Bladder and sexual function following resection for rectal cancer in a randomized clinical trial of laparoscopic versus open technique. Br J Surg. 2005 Sep;92(9):1124-32. doi: 10.1002/bjs.4989. PMID 15997446
- [Background] Maurer CA, Z'Graggen K, Renzulli P, Schilling MK, Netzer P, Buchler MW. Total mesorectal excision preserves male genital function compared with conventional rectal cancer surgery. Br J Surg. 2001 Nov;88(11):1501-5. doi: 10.1046/j.0007-1323.2001.01904.x. PMID 11683749
- [Background] Bouchet-Doumenq C, Lefevre JH, Bennis M, Chafai N, Tiret E, Parc Y. Management of postoperative bladder emptying after proctectomy in men for rectal cancer. A retrospective study of 190 consecutive patients. Int J Colorectal Dis. 2016 Mar;31(3):511-8. doi: 10.1007/s00384-015-2471-8. Epub 2015 Dec 22. PMID 26694925
- [Background] Sethia KK, Selkon JB, Berry AR, Turner CM, Kettlewell MG, Gough MH. Prospective randomized controlled trial of urethral versus suprapubic catheterization. Br J Surg. 1987 Jul;74(7):624-5. doi: 10.1002/bjs.1800740731. PMID 3304522
- [Background] Ratnaval CD, Renwick P, Farouk R, Monson JR, Lee PW. Suprapubic versus transurethral catheterisation of males undergoing pelvic colorectal surgery. Int J Colorectal Dis. 1996;11(4):177-9. doi: 10.1007/s003840050038. PMID 8876274
- [Background] Perrin LC, Penfold C, McLeish A. A prospective randomized controlled trial comparing suprapubic with urethral catheterization in rectal surgery. Aust N Z J Surg. 1997 Aug;67(8):554-6. doi: 10.1111/j.1445-2197.1997.tb02037.x. PMID 9287924
- See also: Southern Medical University, China — http://www.fimmu.com/index_com.html
- See also: Nanfang Hospital, China — http://www.nfyy.com/
- See also: Chinese Anti-Cancer Association — http://www.caca.org.cn/